CLINICAL TRIAL: NCT03284905
Title: Probiotic Intervention for Acute Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Probi AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SP17
Record Dates: First submitted 2017-09-13; First posted 2017-09-15 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Stress

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics (Active Comparator)
  Interventions: Dietary Supplement: Probiotic supplement
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo supplement

INTERVENTIONS:
Dietary Supplement: Probiotic supplement — Capsule containing freeze dried probiotic bacteria together with maize starch
  Arms: Probiotics
Dietary Supplement: Placebo supplement — Capsule containing maize starch
  Arms: Placebo

SUMMARY:
Efficacy of probiotics on acute stress

ELIGIBILITY:
Inclusion Criteria:

* 19-35 years
* SMBQ-score ≥3.75
* Understand Swedish in spoken and written terms
* Willing and able to give written informed consent for participating in the study
* Intake of probiotics within two weeks prior to the start of the study

Exclusion Criteria:

* BMI> 30
* Pregnant
* Antibiotic treatment in the last three months
* Known disease (diabetes, pulmonary or cardiovascular disease, celiac disease, thyroid problems, gastrointestinal disease) or mental illness
* Use of psychotropic drugs, beta blockers, asthma or rheumatoid arthritis drugs, steroid drugs or local steroid treatment

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2018-04-04 (Actual); Study Completion 2018-04-04 (Actual)

PRIMARY OUTCOMES:
Reduction of the cortisol level during acute stress | 2.5 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Food Technology, Engineering and Nutrition, Lund University, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No